CLINICAL TRIAL: NCT03772457
Title: To Explore the Predictive Value of Infarction Volume on Hemorrhagic Transformation in Newly Diagnosed Ischemic Stroke/TIA With Non-valve Atrial Fibrillation(NVAF) Patients Using Rivaroxaban
Brief Title: Predictive Value of Infarction Volume on Hemorrhagic Transformation in Ischemic Stroke/TIA With Non-valve Atrial Fibrillation(NVAF) Patients Using Rivaroxaban
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Bayer (Industry); Taizhou Hospital (Other); Zhuji People's hospital (Unknown); Shaoxing People's Hospital (Other); Jinhua Central Hospital (Other); HaiyanPeople's hospital (Unknown); Wenzhou Central Hospital (Other); The Central Hospital of Lishui City (Other); Dongyang People's Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: InV HT RAF 1010
Record Dates: First submitted 2017-10-10; First posted 2018-12-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cerebrovascular Stroke; Intracranial Hemorrhages; Anticoagulant; Matrix Metalloproteinases
MeSH Terms: conditions — Stroke; Intracranial Hemorrhages | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban — new oral anticoagulant molecules which is the selective factor Xa inhibitor

SUMMARY:
This study was aimed at patients with newly diagnosed stroke / TIA associated with nonvalvular atrial fibrillation. We will observe the effect of early using rivaroxaban anticoagulation on hemorrhagic transformation, and explore the predictive value of multi-mode MRI infarct volume / MMP-9 on hemorrhagic transformation after anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥18;
2. Were newly diagnosed asischemic stroke/TIA concomitant NVAF;
3. Prescribedand accept Rivaroxaban;
4. Sign thewritten informed consent.

Exclusion Criteria:

1. Renal impairment (CrCl<15 ml/min) or severe hepatic impairment.
2. Significant hemorrhagic transformation (parenchymal hematoma type I or type II by the ECASS definition).
3. Stroke or TIA caused by large artery atherosclerosis
4. Planned major surgery or invasive intervention
5. Active internal bleeding
6. Malignancy or other serious medical conditions with a life expectancy <6 months
7. Allergery to Rivaroxaban
8. Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed ischemic stroke/TIA patients with NVAF who sign the informed consent and receiveRivaroxaban treatment in the in-patient ward.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Susceptibility weighted imaging(SWI) detection of newly developed hemorrhagic transformation after 14 days of rivaroxaban treatment | 14 days after enrolling

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China